CLINICAL TRIAL: NCT06317545
Title: Effects of Nirschl Exercises With and Without Mulligan Taping in Lateral Epicondylitis
Brief Title: Effects of Nerchal Exercises on Lateral Epicondylitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AH/23/0167/shan ali
Record Dates: First submitted 2024-01-28; First posted 2024-03-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nirshl exercise with Mulligan Taping (Experimental): This group will be treated with Nirshl exercises with Mulligan taping
  Interventions: Other: Mulligan Taping
- Nirshl exercise without Mulligan taping (No Intervention): This group will be treated with Nirshl exercises only.

INTERVENTIONS:
Other: Mulligan Taping — Mulligan taping involves the application of tape to the lateral aspect of the elbow to offload stress during movement of the extensor tendons.
  Arms: Nirshl exercise with Mulligan Taping

SUMMARY:
Painful condition of lateral epicondyle of the humerus characterized by the inflammation of the tendons during loading of the wrist extensor muscles is a common musculoskeletal presentation in men and women between 35 and 54 years of age. The above symptom is associated with a clinical diagnosis of lateral elbow tendinopathy (LET), also known as tennis elbow or lateral epicondylalgia the two effective treatment approaches for lateral epicondylitis are Nirschl exercises and Mulligan taping. This study aims to evaluate the effectiveness of Nirschl exercises with or without Mulligan taping in treating lateral epicondylitis. The study design for this project employs a randomized controlled trial and a sample of individuals with lateral epicondylitis randomly assigned in one of the two groups i.e., Nirschl exercises only and Nirschl exercises with Mulligan taping. Nirschl exercises involve the eccentric strengthening of the wrist extensor muscles and forearm. The participants in both groups will receive Nirschl exercises while the second group will also receive Mulligan taping, which involves the application of tape to the lateral aspect of the elbow to offload stress during movement of the extensor tendons. Different outcome measures including pain intensity, functional disability, grip strength, range of motion will be evaluated using, PRTEE Scale, Visual Analogue Scale (VAS) and Calibrated Jammer hand held dynamometer. Statistical analysis, including independent t-tests or chi-square tests, will be conducted to compare the outcomes between the two groups. The significance level will be set at p < 0.05. This study will contribute to the evidence base regarding the efficacy of Nirschl exercises and Mulligan taping in managing lateral epicondylitis and will help the clinicians and patients in deciding the best treatment approach for lateral epicondylitis.

ELIGIBILITY:
Inclusion Criteria:

* Pain and tenderness over lateral epicondyle
* at least two out of three tests for the lateral epicondylitis including Cozen's test, Mill's maneuver, or resisted middle finger extension positive

Exclusion Criteria:

* Individuals with a history of recent trauma of upper limbs
* Recent administration of platelet-rich plasma containing growth factors,
* Patients which had taken physical therapy of any sort in the past 6 months
* occupation-related pain were ruled out.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 3 week consist of 6 sessions
  Pain will be measured using Visual Analogue Scale (VAS), min0 and max 10
Grip strength | 3 week consist of 6 sessions
  It will be measured using calibrated Jammer hand-held dynamometer.

SECONDARY OUTCOMES:
Disability | 3 week consist of 6 sessions
  It will be measured using PRTEE scale. 0-10 scale

CONTACTS AND LOCATIONS:
Overall Officials: Sana ullah, MSPT, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - BARKI Advanced Physiotherapy Center, Multan, Punjab Province
  - KAIMS Physiotherapy and Rehabilitation Center, Multan, Punjab Province

IPD SHARING:
Plan to Share IPD: No